CLINICAL TRIAL: NCT03949465
Title: An Open Label Trial of Repetitive Transcranial Magnetic Stimulation (rTMS) for Peri-partum Depression.
Brief Title: rTMS for Peripartum Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment remains at zero.
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB18-1175
Record Dates: First submitted 2019-05-06; First posted 2019-05-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Postpartum Depression; Antepartum Depression; Peripartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Open label iTBS rTMS (Experimental): Participants will receive repetitive transcranial magnetic stimulation (rTMS) as a treatment for depression
  Interventions: Device: Transcranial Magnetic Stimulator

INTERVENTIONS:
Device: Transcranial Magnetic Stimulator — Repetitive Transcranial magnetic stimulation (rTMS) will be delivered using a MagPro X100 device with B70 coil and the intermittent theta burst (iTBS) protocol to the left dorsolateral prefrontal cortex. Participants will receive daily treatments (Monday-Friday) over four weeks

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a neuromodulatory technique that is effective in major depression. There is preliminary evidence suggesting that rTMS is effective in peripartum depression as well, however this comes from a number of very small studies.

The objective is to study the effectiveness of rTMS in peripartum depression. The investigators will do so using an open label design in which participants will receive rTMS for four weeks. The focus is on clinical improvement in depressive symptoms; however the investigators will also look at other aspects such as perinatal anxiety and maternal-infant bonding as measured by self-report questionnaires.

DETAILED DESCRIPTION:
Peripartum Depression (PPD) is common and severely disabling. Pharmacological intervention remains the first line of treatment, however many patients do not experience any benefits from them. Furthermore, many women are hesitant about pharmaceutical interventions due to the unknown effects on foetal health and lactation. Hence novel treatment approaches are required for such patients. Neuromodulation techniques involve selective targeting of brain areas which are promising avenues for such depressed patients.

Transcranial magnetic stimulation (rTMS) is an investigational and therapeutic modality that impacts neurons by delivering patterned energy safely and noninvasively. In response to this patterned energy, neurons fire, and adapt by changing their connection strengths. This change in connection strength is believed to be the underlying mechanism whereby rTMS has therapeutic benefit in conditions such as Major Depressive Disorder (MDD). There are preliminary evidences suggesting that it is effective in PPD as well, however this comes from a number of very small studies and is therefore unclear.

Given the promising preliminary evidence, the investigators propose to study the effectiveness of intermittent Theta-Burst Stimulation rTMS (iTBS) to the left dorsolateral prefrontal cortex (DLPFC) in treating PPD. Participants with PPD will receive iTBS rTMS for four weeks (20 sessions) in an open label manner. The primary measure will be clinical improvement in depressive symptoms as measured by change in the Montgomery-Asberg Depression Rating Scale (MADRS) with iTBS-rTMS. In addition, the investigators will look at other aspects such as peripartum anxiety and maternal attachment during treatment and 8 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Women currently experiencing peripartum depression as determined by the MINI-International Neuropsychiatric Interview
* Depressive episode of at least moderate severity, as indicated by a score of ≥15 (ante-partum) or ≥12 (post-partum) on the Edinburgh Post-Natal Depression Scale (EPNDS).
* Are currently pregnant or 1 month post-delivery
* Refuse antidepressant therapy, or have depression that has not improved with psychotropics and/or psychotherapy
* Be willing to remain on a stable medication regimen for 2 weeks prior the study and during the study
* Aged 18-40 years

Exclusion Criteria:

* Epilepsy, history of seizures or pre-eclampsia
* Previous Stroke
* Current Alcohol Use Disorder
* History of psychosis
* Bipolar Disorder
* Current suicidal ideation
* Intracranial metallic objects (dental hardware is not an exclusionary criteria)
* Unstable medical condition
* have failed a course of ECT in the current episode. Previous ECT treatment outside of the current episode does not influence inclusion.
* history of non-response to rTMS treatment .
* have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of epilepsy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
* have concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* have any significant obstetrical complications
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
* have a clinically significant laboratory abnormality, in the opinion of study physician
* are currently (or in the last 4 weeks) taking lorazepam greater than 2 mg daily (or equivalent) due to the potential to limit rTMS efficacy
* are currently (or in the last 4 weeks) taking lorazepam greater than or equal to 2 mg daily

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4).
  Change from baseline in severity of depressive symptoms at 2 weeks and 4 weeks as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.

SECONDARY OUTCOMES:
Rate of Clinical Remission of Depressive Symptoms | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  Number of participants with a score of </= 10 on the MADRS
Rate of Clinical Response in Depressive Symptoms | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  Number of participants with a >/= 50% reduction in MADRS scores
Perinatal Anxiety Symptoms | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  Perinatal Anxiety symptoms will be assessed using the Perinatal Anxiety Screening Scale (PASS). The PASS measures self-reported feelings of anxiety in the peripartum period. PASS scores range from 0-93, interpretations are as follows: 0-20 = asymptomatic, 21-41 = mild-moderate symptoms, and 42-93 = severe symptoms.
Anxiety Symptoms | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  The State-Trait Anxiety Inventory (STAI) measures self reported feelings of extrinsic "state" anxiety and intrinsic "trait" anxiety. The STAI scores range from 20-80, with higher scores correlating to greater anxiety.
Antenatal Maternal Attachment | If the participant is antenatal, the MAAS will be administered at baseline and after rTMS treatment (week 4).
  The Maternal Antenatal Attachment Scale (MAAS) assesses self-reported feelings of the mother-child relationship before birth. Scores range from 19-95 on the MAAS, with lower scores representing lower levels of attachment.
Postnatal Maternal Attachment | If the participant is postnatal, the scale will be administered at baseline and after rTMS treatment (week 4). All participants will complete the MPAS at 8 weeks postpartum.
  The Maternal Postnatal Attachment Scale (MPAS) assesses self-reported feelings of the mother-child relationship after birth. Scores range from16-80 on the MPAS, with lower scores representing lower levels of attachment.
Quick Inventory of Depressive Symptomatology- Self-report (QIDS-SR) | Administered at baseline, halfway (week 2) and after rTMS treatment (week 4). All participants will complete the QIDS-SR at 8 weeks postpartum.
  The QIDS -SR is a self-reported measure of depressive symptoms. Total scores range from 0 to 27, with higher scores representing greater severity of depression. Score interpretations are as follows: 0-7 = normal, 8-12 = mild, 13-16 = moderate, 17-20 = moderate to severe, 21-27 = severe.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Daily Monday-Friday throughout study (4 weeks)
  Adverse events will be tracked and recorded
Side Effects | Daily Monday-Friday throughout study (4 weeks)
  Side effects will be tracked through a comfort rating questionnaire. The comfort rating questionnaire assesses the frequency and severity of side effects common to rTMS treatment. Severity of individual side effects are rated from 1 (none) to 10 (extreme).
Toronto Side Effects Scale (1 week) (TSES) | Administered at baseline, halfway (week 2) and after rTMS treatment (week 4).
  The Toronto Side Effects Scale measures frequency and severity of a variety of side effects over the past week. Frequency and severity of each symptom are rated on a scale of 1 - 5, with higher scores corresponding to more frequent/severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided